CLINICAL TRIAL: NCT05786378
Title: Assessment of The Efficacy of Intratympanic Platelet Rich Plasma for Treatment of Sensorineural Hearing Loss.
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mahmoud Hassan Ali, Resident doctor at Otolaryngology Departement, Principal Investigator, Assiut University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Intratympanic PRP
Record Dates: First submitted 2023-03-07; First posted 2023-03-27 (Actual); Last update posted 2023-04-19 (Actual); Status verified 2023-04

CONDITIONS: Hearing Loss, Sudden; Hearing Loss, Sensorineural; Hearing Loss
MeSH Terms: conditions — Hearing Loss, Sudden; Hearing Loss, Sensorineural; Hearing Loss | interventions — Anesthesia, Local; Injection, Intratympanic

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- platlet rich plasma (Experimental)
  Interventions: Biological: Platelet Rich Plasma; Drug: local anesthesia in external auditory canal; Procedure: Intratympanic Injection

INTERVENTIONS:
Biological: Platelet Rich Plasma — Sample of patient's blood drawn at time of Treatment; the blood drawing occurs with addition of anticoagulant such as citrate dextrose A to prevent platelet activation prior to its use.
  Obtain whole blood by venipuncture in acid citrate dextrose (ACD) tubes. Centrifuge the blood using a 'soft' spin. Transfer the supernatant plasma containing platelets into another sterile tube (without anticoagulant).
  Centrifuge tube at a higher speed (a hard spin) to obtain a platelet concentrate.
  The lower 1/3rd is PRP and upper 2/3rd is platelet-poor plasma (PPP). At the bottom of the tube, platelet pellets are formed.
  PRP activation prior to injection. PRP can be activated exogenously by calcium chloride.
Drug: local anesthesia in external auditory canal — local anesthesia cream (lidocaine cream) will be applied in external auditory canal for 15 minutes
Procedure: Intratympanic Injection — 0.5-1 ml of PRP will be injected in middle ear cavity in round window niche Using microscope or endoscope.

SUMMARY:
Assessment of the efficacy of Intratympanic platelet rich plasma injection for treatment of idiopathic suden sensorineural hearing loss

DETAILED DESCRIPTION:
Sensorineural hearing loss is the collective term for hearing damage to the cochlea and auditory nerve and is by far the most common type of hearing loss in adults, accounting for over 90% of all cases. Sensorineural hearing loss is a heterogeneous disorder, which can arise due to damage to pathway for sound impulses from the hair cells of inner ear to auditory nerve and less commonly brain.

Sensorineural hearing loss is a challenge to physicians, as it progresses with age and causes significant reductions in quality of life and there are no treatments to reverse its effects, other than sound amplification with the use of hearing aids or direct auditory nerve stimulation via cochlear implantation.

Platelet-rich Plasma (PRP) Therapy is a cutting-edge procedure that is revolutionizing the hearing loss and deafness. Intratympanic instillation of Platelet-rich Plasma (PRP) does wonder to the hair cells of inner ear, thus improving the hearing.

ELIGIBILITY:
Inclusion Criteria:

* Patients have sudden idiopathic sensorineural hearing loss

Exclusion Criteria:

1. patients has previous ear surgery.
2. patients has absent cochlea in CT or MRI
3. patients has Cancer,Chronic liver disease, Hemodynamic instability,Hypofibrinogenemia, Platelet dysfunction syndromes, Systemic disorder, sepsis, Low platelet count.

Ages: 5 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 23 (Estimated)
Dates: Start 2023-06-01 (Estimated); Primary Completion 2024-01 (Estimated); Study Completion 2024-02 (Estimated)

PRIMARY OUTCOMES:
Changes in Pure Tone Averages | 6 weeks
  Continuous pure tone averages calculated from pure tone audiometry will be summarized using the mean, standard deviation, median, 25th percentile, 75th percentile, minimum and maximum.

CONTACTS AND LOCATIONS:
Locations (1):
- Otorhinolaryngeology Departement, Faculty of Medicine , Assuit Univerisity, Asyut, Assuit, Egypt